CLINICAL TRIAL: NCT02128308
Title: A Open-label, Single Sequence Clinical Trial to Investigate the Pharmacokinetic Characteristics of Second-Line Anti-Tuberculosis Agents After Multiple Oral/Intramuscular Administration in Healthy Male Volunteers
Brief Title: Clinical Trial to Investigate the Pharmacokinetics of Second-Line Anti-Tuberculosis Agents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jae Yong Chung, Assistant Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBPK
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Antituberculosis agents; Pharmacokinetics
MeSH Terms: interventions — Levofloxacin; Cycloserine; Aminosalicylic Acid; Prothionamide; Pyrazinamide; Moxifloxacin; Kanamycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levofloxacin and Streptomycin added (Experimental): Levofloxacin and Streptomycin added : Cycloserine(CS) 250mg bid, P-aminosalicylic acid(PAS) 2 pack bid, Prothionamide(PTH) 250mg (125mg x 2 tab) bid, Pyrazinamide(PZA) 1500mg (500mg x 3 tab) qd, Levofloxacin 750mg (500mg x 1.5 tab) qd, Streptomycin 1g IM qd
  Interventions: Drug: Levofloxacin and Streptomycin added
- Moxifloxacin and Kanamycin added (Experimental): Cycloserine(CS) 250mg bid, P-aminosalicylic acid(PAS) 2 pack bid, Prothionamide(PTH) 250mg (125mg x 2 tab) bid, Pyrazinamide(PZA) 1500mg (500mg x 3 tab) qd, Moxifloxacin 400mg (400mg x 1 tab) qd, Kanamycin 1g IM qd
  Interventions: Drug: Moxifloxacin and Kanamycin added

INTERVENTIONS:
Drug: Levofloxacin and Streptomycin added
  Other Names: Cycloserine; P-aminosalicylic acid; Prothionamide; Pyrazinamide; levofloxacin; steptomycin
  Arms: Levofloxacin and Streptomycin added
Drug: Moxifloxacin and Kanamycin added
  Other Names: Cycloserine; P-aminosalicylic acid; Prothionamide; Pyrazinamide; moxifloxacin; kanamycin
  Arms: Moxifloxacin and Kanamycin added

SUMMARY:
This study aims to investigate the pharmacokinetic characteristics of second-line anti-tuberculosis agents after oral/intramuscular administration in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subject aged 20 to 50 at screening
* a body weight in the range of 55 kg (inclusive) to 90 kg (inclusive) with ideal body weight range of 19.0 to 26.0 subjects who decide to participate voluntarily and write a informed consent form

Exclusion Criteria:

* subjects who have clinically significant disease of cardiovascular, respiratory, renal, endocrinological, hematological, gastrointestinal, neurological(central nervous system), psychiatric disorders or malignant tumor
* subject judged not eligible for study participation by investigator.

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-11; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
AUC (area under the plasma concentration-time curve) | Predose and 2d 0h, 3d 0h, 4d 0h, and 5d 0, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24h postdose
  AUC (Area under the plasma concentration versus time curve), Cmax(maximum plasma concentration)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park SI, Oh J, Jang K, Yoon J, Moon SJ, Park JS, Lee JH, Song J, Jang IJ, Yu KS, Chung JY. Pharmacokinetics of Second-Line Antituberculosis Drugs after Multiple Administrations in Healthy Volunteers. Antimicrob Agents Chemother. 2015 Aug;59(8):4429-35. doi: 10.1128/AAC.00354-15. Epub 2015 May 18. PMID 25987620